CLINICAL TRIAL: NCT04315831
Title: Safety and Effectiveness of Transdermal Buprenorphine in Cancer Pain: an Observational Study (SOOTHE)
Brief Title: Safety and Effectiveness of Transdermal Buprenorphine in Cancer Pain
Acronym: SOOTHE
Status: Completed | Type: Observational
Sponsor: Taiwan Mundipharma Pharmaceuticals Ltd. (Industry)
Collaborators: Chang Gung Memorial Hospital (Other); Changhua Christian Hospital (Other); Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BUP17-TW-401
Record Dates: First submitted 2020-03-16; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Cancer
Keywords: Transdermal Buprenorphine, Cancer pain, QOL, NRS, Narcotics
MeSH Terms: conditions — Neoplasms; Cancer Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Transdermal Buprenorphine — Intervention will be applied for patients with moderate to severe cancer pain
  Other Names: no other intervention

SUMMARY:
Buprenorphine transdermal patch is newly available in Taiwan in June 2017, the trade name is Transtec, and the available dosages are 35 μg/h and 52.5 μg/h. Taiwan is the first Asia country which launched Transtec for cancer pain treatment. Although the efficacy of transdermal buprenorphine has been demonstrated in some randomized, placebo-controlled studies and also conducted a large scale post-marketing surveillance study in Germany, therefore the local scientific data is required for Asia experience. Due to above rationale, this observational study will be initiated in Taiwan, to build up the first real-world scientific data in Asia.

The objective of this study is to collect the safety and effectiveness of transdermal buprenorphine in routine clinical practice, in particular, to collect data in population with controlled cancer pain and stable titration from previous opioid analgesics in Taiwan.

DETAILED DESCRIPTION:
The objective of this observational study is to collect effectiveness and safety data on the labelled use of buprenorphine transdermal patches (Transtec 35 μg/h and 52.5 μg/h) under regular and routine clinical conditions in Taiwan for cancer patients with moderate to severe cancer pain (NRS Score>=4) and strong opioids are needed for their pain treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients aged 20 years old and over
2. ECOG <3
3. Moderate or severe pain intensity with stable titration from previous opioid analgesics, 7 days at least prior to enrolment and with the dose equivalent to oral morphine ranging from 60 to 120 mg/day in previous treatment
4. Cancer-related pain that requires treatment with continuous around-the-clock strong opioid analgesic
5. Patients who are going to start Transtec treatment per clinical judgment, according to the locally approved labeling, are eligible.
6. Patients who are able to communicate and fill out the questionnaire forms
7. Patient provided signed informed consent

Exclusion Criteria:

1. Patients diagnosed with non-cancer pain or unexplained pain
2. Patients who have constipation (CTCAE grade 3 and above)
3. Patients with uncontrolled or unstable cardiac disease
4. Abnormal lab results, with obvious clinical significance, such as ALT or AST>= 3 fold of upper limit of normal value or liver function of Child C grade prior to study
5. ALT or AST >= 5 fold of upper limit of normal value for patients with liver metastasis or primary liver cancer
6. Pregnant or nursing (lactating) women
7. Patients who are drug or alcohol abuse
8. Patients who have hypersensitivity to buprenorphine
9. Patients who are clinically unstable or have a life expectancy of less than 8 weeks making completion of the trial unlikely
10. With any contraindications or using prohibited medication per locally approved

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caner patients with moderate to severe cancer pain
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Adverse drug reaction | Week 3 to Week 4 or early termination
  Number and percentage of patients with adverse drug reactions and serious adverse drug reactions

SECONDARY OUTCOMES:
Pain intensity and interference | whole study-1 month
  Pain intensity and interference measured by the Brief Pain Inventory (BPI)
Daily pain intensity measured by a numerical rating scale (NRS) by patients | 1 month
  Daily pain intensity measured by a numerical rating scale (NRS) designed in a patient diary card
Quality of life of the patients | 1 month
  Quality of life measured by the EORTC QLQ-C30
Quality of sleep of the patients | 1 month
  Quality of sleep measured by a NRS
Number of breakthrough pain | 1 month
  Number of breakthrough pain during the observational period
Treatment discontinuation and associated reasons | during study period-1 month
  reason for stop treatments

OTHER OUTCOMES:
ECG changes | 1 month of study period
  The change from baseline in ECG measurement at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Shi Chen, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital- Linko Branch, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
No plan to share the individual participant data to other researchers unless formal request been reviewed and pproval

REFERENCES:
- [Derived] Huang TL, Huang YM, Hou MM, Lu CH, Chao TY, Chiu TJ, Chang YS, Lin SH, Lin CH, Chen YH, Wang CH, Chen JS, Shen WC. Safety and effectiveness of transdermal buprenorphine in cancer pain: An observational study in Taiwan (SOOTHE). Asia Pac J Clin Oncol. 2023 Apr;19(2):e45-e53. doi: 10.1111/ajco.13772. Epub 2022 May 22. PMID 35604203
- [Derived] Shen WC, Hou MM, Huang TL, Wang CH, Huang YM, Chen JS, Chen ML. Transdermal buprenorphine improves overall quality of life and symptom severity in cancer patients with pain. J Clin Nurs. 2023 Feb;32(3-4):539-547. doi: 10.1111/jocn.16303. Epub 2022 Mar 31. PMID 35362192